CLINICAL TRIAL: NCT01885806
Title: Repetitive Transcranial Magnetic Stimulation for Apathy Treatment in Alzheimer's Disease: a Randomised, Double-blind, Controlled Study
Brief Title: Repetitive Transcranial Magnetic Stimulation for Apathy Treatment in Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Breno Satler de Oliveira Diniz, Assistant Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE: 15388913.6.0000.5149
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Alzheimer's Disease; Apathy
Keywords: Apathy; Alzheimer's disease; Cognition; Burden of Care
MeSH Terms: conditions — Alzheimer Disease; Lethargy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Repetitive TMS (Experimental): Patients will receive 10 consecutive sessions of repetitive transcranial magnetic stimulation with the following protocol:
  Frequency: 10 Hz Intensity: 90% motor limiar Session duration: 16 minutes (20 sequencies of 6 seconds of stimulation followed by intervals of 30 seconds); Localization: Left pre-frontal dorsolateral cortex;
  Interventions: Device: Magnetic Stimulator Magstim Rapid 2
- Sham TMS (Sham Comparator): Patients will receive 10 consecutive sessions of sham transcranial magnetic stimulation following the same protocol as the intervention arm, but with no magnetic stimulation of the brain.
  Interventions: Device: Sham Magnetic Stimulator

INTERVENTIONS:
Device: Magnetic Stimulator Magstim Rapid 2 — All procedures will use the Magnetic Stimulator Magstim Rapid 2. Total of session: 10 rTMS protocol: Freqüency: 10 Hz Intensity: 90% limiar motor Session duration: 16 minutes (20 TMS sequences of 6 second with intervals of 30 seconds between each sequence) Location: Left dorsolateral pre-frontal cortex
  Other Names: rTMS
  Arms: Repetitive TMS
Device: Sham Magnetic Stimulator — This intervention will follow the same protocol of the rTMS except that subjects will not receive magnetic stimulation of the brain.
  Total of session: 10
  Other Names: Sham
  Arms: Sham TMS

SUMMARY:
We aim to evaluate the safety and efficacy of repetitive transcranial magnetic stimulation (rTMS) for apathy treatment in patients with Alzheimer's disease (AD). We hypothesize that rTMS will be superior to placebo to reduce apathy symptoms and severity in patients with AD.

DETAILED DESCRIPTION:
This study aims to enroll 40 patients with mild and moderate Alzheimer's disease with apathy symptoms that will be randomized to receive rTMS or sham procedure. Subjects will be randomized in two arms (rTMS or sham procedure) in 1:1 proportion.

Eligibility criteria:

* Diagnosis of Alzheimer's disease, mild and moderate stage (MMSE range from 10 to 20);
* Diagnosis of apathy;
* age between 60 and 85 years-old;
* On stable doses of cholinesterase inhibitors (donepezil, rivastigmine, galantamine) or memantine for at least 6 months prior to enrollment;

The primary outcome measures is the Apathy Inventoire. Secondary outcome measures are the NPI score, ADAS-cog scores and the Zarit Burden Scale scores.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60 to 85 years-old
* Mild or moderate Alzheimer's disease (MMSE scores between 10 and 20)
* Apathy diagnosis
* On stable doses of cholinesterase inhibitors (donepezil, galantamine, rivastigmine) and/or memantine for at least 6 months prior to enrollment

Exclusion Criteria:

* history of epilepsy or convulsions
* History of migraine or headaches episodes twice per week or more
* History of neurodegenerative diseases other than Alzheimer's disease
* Current use of first generation antipsychotics, clozapine, tricyclic drugs or anticonvulsants
* History of cerebral ischemic episode

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in apathy symptoms | 12 weeks
  Reduction of 30% in the Apathy Inventoire scores between baseline and 12 weeks after treatment.

SECONDARY OUTCOMES:
Change in ADAS-Cog scores | 12 weeks
  Improvement in ADAS-Cog scores between baseline and 12 weeks after treatment.
Change in the Zarit Burden Scale | 12 weeks
  Reduction in the Zarit Burden Scale between baseline and 12 weeks after treatment.

OTHER OUTCOMES:
Safety assessment | 4th week, 8th week, 12th week
  Assessment of rTMS safety by the UKU scale.

CONTACTS AND LOCATIONS:
Overall Officials: Breno S Diniz, MD, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Outside of U.S., Brazil